CLINICAL TRIAL: NCT06597032
Title: The Resilience Challenge: FERN (Fostering Emotional Resilience During a Time of National Stress)
Brief Title: The Resilience Challenge: Fostering Emotional Resilience During a Time of National Stress
Acronym: FERN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor of Medical Social Sciences, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00222090
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Stress; Positive Affect
Keywords: Positive Affect; Resilience Challenge; Positive Psychology; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resilience Challenge (Experimental): The Resilience Challenge Study is an online program containing a series of positive emotion skills for individuals experiencing stress and distress during their everyday life. The online program specifically targets positive emotion and offers an array of skills in a self-guided online delivery platform. Participants will, over the course of 6-8 weeks, access weekly skill lessons, daily homework, and daily emotion reporting. The skill lessons will include: positive events, savoring, gratitude, everyday mindfulness, mindfulness meditation, positive reappraisal, self-compassion, personal strengths, and attainable goals.
  Interventions: Behavioral: Resilience Challenge

INTERVENTIONS:
Behavioral: Resilience Challenge — We previously have tested this online program in people facing health- and work-related stressors (e.g., dementia caregivers, healthcare workers), and in 2020 we enrolled adults in a test of the online program to support coping with the stress of the COVID pandemic. This intervention has been tailored for a widespread, public audience (e.g., we have added a few other safety measures including limits on public forum posting and have clarified wording on some of the intervention content to make it clearer and easier to understand).

SUMMARY:
The goal of this clinical trial is to examine the effects of an online positive psychological intervention on positive emotion, anxiety, depression, feelings of social isolation, sleep disturbance and a sense of meaning and purpose in the general public. The main question it aims to answer is:

Will the practice of positive emotion skills via a self-guided online platform reduce feelings of anxiety, depression, social isolation, and sleep disturbance, as well as increase well-being, positive emotion, a sense of meaning and purpose, life satisfaction, and general self-efficacy?

Participants will take part in an online positive psychological skill learning intervention for 6-8 weeks. Prior to beginning, immediately after, and 4 weeks after, participants will fill out measures of their wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, Access to device connected to the internet

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11659 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
PROMIS Positive Affect CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later

SECONDARY OUTCOMES:
PROMIS Depression CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later
PROMIS Anxiety CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later
PROMIS Meaning and Purpose CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later
PROMIS Social Isolation CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later
PROMIS Sleep Disturbance CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later
PROMIS General Self-Efficacy CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later
PROMIS General Life Satisfaction CAT | At baseline, after completion of 6-8 week intervention, and 4 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Judith T Moskowitz, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States